CLINICAL TRIAL: NCT06580574
Title: Sintilimab With Selective Combination of Sintilimab, IBI310 and Lenvatinib Used for Organ Preservation in Non-metastatic Gastric or Colon Cancers With Mismatch Repair Deficiency or High Microsatellite Instability
Brief Title: Immune Checkpoint Inhibitors for Organ Preservation in Non-metastatic dMMR/MSI-H Gastric or Colon Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG-IMAGINE-06
Record Dates: First submitted 2024-08-24; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Colon Cancer; MSI-H; DMMR Cancer
Keywords: Organ preservation; immunotherapy; anti-VEGF
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dMMR/MSI-H gastric cancer (Experimental): PD1/PDL1 antibody monotherapy will be given per local treatment standards.
  If (near-) clinical complete response is not achieved after 24 weeks of PD1/PDL1 antibody monotherapy, then combination of intensive immunotherapy plus anti-VEGF treatment will be used.
  If (near-) clinical complete response is not achieved after 24 weeks of intensive immunotherapy plus anti-VEGF treatment, radical surgery will be recommended.
  Interventions: Drug: PD1/PDL1 antibody monotherapy, up to 24 weeks; Combination Product: Intensive immunotherapy plus anti-VEGF treatment, up to 24 weeks; Procedure: Radical surgery
- dMMR/MSI-H colon cancer (Experimental): PD1/PDL1 antibody monotherapy will be given per local treatment standards.
  If (near-) clinical complete response is not achieved after 24 weeks of PD1/PDL1 antibody monotherapy, then combination of intensive immunotherapy plus anti-VEGF treatment will be used.
  If (near-) clinical complete response is not achieved after 24 weeks of intensive immunotherapy plus anti-VEGF treatment, radical surgery will be recommended.
  Interventions: Drug: PD1/PDL1 antibody monotherapy, up to 24 weeks; Combination Product: Intensive immunotherapy plus anti-VEGF treatment, up to 24 weeks; Procedure: Radical surgery

INTERVENTIONS:
Drug: PD1/PDL1 antibody monotherapy, up to 24 weeks — non-specific, according to Drug Instructions
Combination Product: Intensive immunotherapy plus anti-VEGF treatment, up to 24 weeks — Sintilimab 200mg, ivgtt, q21d; IBI310 1mg/kg, ivgtt, q42d; Lenvatinib 8mg (starting from 4mg), po, qd
Procedure: Radical surgery — Radical surgery will be recommended per local treatment standards.

SUMMARY:
This study intends to explore the role of PD1/PDL1 antibody with selective combination of Sintilimab, IBI310 and Lenvatinib in organ preservation in non-metastatic dMMR/MSI-H gastric or colon cancers with mismatch repair deficiency or high microsatellite instability

ELIGIBILITY:
Inclusion Criteria:

* Subjects are able to comprehend the informed consent form, and voluntarily sign the informed consent form.
* Subjects are ≥18 years old on the day of signing the informed consent form, with no gender restrictions.
* Histologically confirmed gastric cancer or colon cancer, without distant metastasis based on CR or MR.
* ECOG performance status of 0-2.
* dMMR confirmed by immunohistochemistry or MSI-H confirmed by PCR and NGS. If MSI status and MMR status were not consistent, whether to enroll this patient should be determine by investigators. Patients with MMR heterogeneity in tumors could not be included.
* Patients who are about to receive or are receiving 24 weeks of PD1/PDL1 antibody monothearpy and have not had the first efficacy assessment.
* Archived tumor tissue samples or freshly obtained tumor tissue samples are available.
* Female subjects of childbearing potential or male subjects with partners of childbearing potential agree to use highly effective contraception from 7 days before the first dose until 120 days after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose.
* Subjects have the ability and willingness to comply with the study protocol's visits, treatment plan, laboratory tests, and other study-related procedures.
* For patients who are about to receive combination of Sintilimab, IBI310 and Lenvatinib. subjects should have good organ function within the first 7 days of initial dosing: HGB ≥ 80g/L, NEU ≥ 1.0*10^9/L, PLT ≥ 75*10^9/L, Cr≤1.5×ULN or CrCl≥50mL/min（Cockcroft-Gault method), TBiL ≤ 1.5×ULN, ALT and AST ≤3 ×ULN; urine protein <2+; if urine protein ≥ 2+, 24 hour urinary protein quantity <2g; INR, APTT, PT ≤ 1.5 ×ULN

Exclusion Criteria:

* Distant metastasis;
* Previous treatment including CTLA4 blockade;
* Subjects with interstitial lung disease or a history of non-infectious pneumonia requiring oral or intravenous corticosteroid treatment.
* Subjects with active autoimmune diseases requiring systemic treatment before the start of the study or those considered at risk of recurrence or planned treatment for autoimmune diseases as judged by the investigator. Except for these conditions: a) skin diseases that do not require systemic treatment (e.g., vitiligo, alopecia, psoriasis, or eczema); b) hypothyroidism caused by autoimmune thyroiditis, requiring stable doses of hormone replacement therapy; c) type 1 diabetes requiring stable doses of insulin replacement therapy; d) childhood asthma fully resolved with no need for intervention in adulthood; e) the investigator judges that the disease will not relapse without external triggering factors.
* Subjects with a history of other malignant tumors within 5 years, excluding cured skin squamous cell carcinoma, basal cell carcinoma, non-invasive bladder carcinoma, localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6, and prostate-specific antigen (PSA) ≤10 ng/mL (if measured) in patients who have undergone curative treatment and have no biochemical recurrence of prostate-specific antigen (PSA)), in situ cervical/breast carcinoma, or Lynch syndrome.
* Subjects with uncontrolled comorbidities, including but not limited to: a) active HBV or HCV infection; b) subjects who are HBsAg positive and/or HCV antibody positive during screening must undergo HBV DNA and/or HCV RNA testing. Only subjects with HBV DNA ≤500 IU/mL (or ≤2000 copies/mL) and/or HCV RNA negative can be enrolled; HBV DNA monitoring will be at the discretion of the investigator based on the subject's condition during the trial; c) known HIV infection or AIDS history; d) active tuberculosis; e) uncontrolled hypertension (resting blood pressure ≥160/100 mmHg), symptomatic congestive heart failure (NYHA II-IV), unstable angina or myocardial infarction within 6 months, or the presence of QTc prolongation or the risk of arrhythmia (baseline QTc >470 msec <Fridericia method correction>, refractory hypokalemia, long QT syndrome, atrial fibrillation with resting heart rate >100 bpm, or severe valvular heart disease); f) active bleeding that cannot be controlled after medical treatment.
* History of allogeneic bone marrow or organ transplantation.
* Previous history of allergic reactions, hypersensitivity reactions, or intolerance to antibody drugs (e.g., severe allergic reactions, immune-mediated hepatotoxicity, immune-mediated thrombocytopenia, or anemia).
* Pregnant and/or lactating females.
* For patients who are about to receive combination of Sintilimab, IBI310 and Lenvatinib: a) Subjects with a history of gastrointestinal perforation or fistula within 6 months before the first dose. If the perforation or fistula has been treated with resection or repair, and the disease is judged to be recovered or improved by the investigator, then enrollment is allowed. b) Subjects who have undergone major surgery within 28 days before the first dose (e.g., major abdominal or thoracic surgery; excluding drainage, diagnostic puncture, or peripheral vascular access replacement). c) Subjects who require systemic corticosteroids (≥10 mg/day prednisone or equivalent) or immunosuppressive therapy for a continuous 7-day period within 14 days before the first dose. Inhaled or locally applied steroids and physiological replacement doses of steroids due to adrenal insufficiency are allowed. Short-term (≤7 days) corticosteroids for prophylaxis (e.g., contrast dye allergy) or treatment of non-autoimmune diseases (e.g., delayed hypersensitivity reaction caused by exposure to allergens) are allowed. d) Toxicity from previous antitumor treatments has not recovered to Grade ≤2 (NCI-CTCAE v5.0) or baseline, except for alopecia, skin pigmentation (allowed at any level), and immune-related adverse reactions requiring physiological replacement (e.g., hypothyroidism, hypopituitarism, type 1 diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Organ preservation rate | The status of cCR or near-cCR and the possibility of organ preservation will be evaluated after completion of PD1/PDL1 antibody monotherapy, 12 weeks after Sintilimab, IBI310 and Lenvatinib, and 24 weeks after Sintilimab, IBI310 and Lenvatinib
  The rate of patients who achieved cCR or near-cCR and did not undergo surgery after completion of established therapy, assessed among all patients who completed established therapy.

SECONDARY OUTCOMES:
Organ preservation rate after completion of PD1/PDL1 antibody monotherapy | The status of cCR or near-cCR and the possibility of organ preservation will be evaluated after completion of PD1/PDL1 antibody monotherapy, an average of 24 weeks
  The rate of patients who achieve cCR or near-cCR and do not undergo surgery after completion of PD1/PDL1 antibody monotherapy, assessed among all patients who completed PD1/PDL1 antibody monotherapy
Organ preservation rate after completion of selective combination of Sintilimab, IBI310 and Lenvatinib | The status of cCR or near-cCR and the possibility of organ preservation will be evaluated 12 weeks and 24 weeks after Sintilimab, IBI310 and Lenvatinib
  The rate of patients who achieved cCR or near-cCR and did not undergo surgery after completion of selective combination of Sintilimab, IBI310 and Lenvatinib, assessed among all patients who do not achieve cCR or near-cCR after PD1/PDL1 antibody monotherapy, and all patients who achieve cCR or near-cCR after PD1/PDL1 antibody monotherapy but have disease progression during follow-up
Objective response rate of selective combination of Sintilimab, IBI310 and Lenvatinib | Baseline up to withdrawal of consent, progressive disease, unacceptable toxicity, or surgery (whichever occurs first), up to 8 years
  Objective response rate (defined as CR+PR) will be reported based on investigator's evaluation according to RECIST 1.1
Disease control rate of selective combination of Sintilimab, IBI310 and Lenvatinib | Baseline up to withdrawal of consent, progressive disease, unacceptable toxicity, or surgery (whichever occurs first), up to 8 years
  Disease control rate (defined as CR+PR+SD) will be reported based on investigator's evaluation according to RECIST 1.1
3 year organ preservation rate | From first dose of PD1/PDL1 antibody until the date of surgery, assessed up to 3 years
  Rate of 3 year surgery-free survival
3 year disease free survival rate | From first dose of PD1/PDL1 antibody until disease progression (local or distant), secondary tumor or death (whichever occurs first), assessed up to 3 years
  Rate of 3 year disease free survival
3 year overall survival rate | From first dose of PD1/PDL1 antibody until death, assessed up to 3 years
  Rate of 3 year overall survival
5 year overall survival rate | From first dose of PD1/PDL1 antibody until death, assessed up to 5 years
  Rate of 5 year overall survival
3 year local recurrence free survival rate | From first dose of PD1/PDL1 antibody until first local failure or death (whichever occurs first), assessed up to 3 years
  Rate of 3 year local recurrence free survival
3 year distant metastasis free survival rate | From first dose of PD1/PDL1 antibody until distant metastasis or death (whichever occurs first), assessed up to 3 years
  Rate of 3 year distant metastasis free survival
3 year surgery free survival rate | From first dose of PD1/PDL1 antibody until radical surgery or death (whichever occurs first), assessed up to 3 years
  Rate of 3 year surgery free survival
Treatment-related adverse event of combination of Sintilimab, IBI310 and Lenvatinib | From first dose of Sintilimab, IBI310 and Lenvatinib to 30 days after last dose of treatment.
  A treatment-related adverse event (TRAE) is defined as any adverse event not present prior to the initiation of drug treatment or any adverse event already present that worsens in intensity or frequency following exposure to the drug treatment. TRAEs were graded using National Cancer Institute (NCI)-CTCAE version 5.0.
Quality of life of combination of Sintilimab, IBI310 and Lenvatinib for gastric cancer patients | From first dose of PD1/PDL1 antibody until death, assessed up to 8 years
  Quality of life will be evaluated using EORTC QLQ-C30 and QLQ-STO22.
Quality of life of combination of Sintilimab, IBI310 and Lenvatinib for colon cancer patients | From first dose of PD1/PDL1 antibody until death, assessed up to 8 years
  Quality of life will be evaluated using EORTC QLQ-C30 and EORTC QLQ-CR29.
Rate of complications | From 7 days before surgery to 12 days after surgey
  Rate of complications in perioperative period
Rate of mortality | From 7 days before surgery to 12 days after surgey
  Rate of mortality in perioperative period

OTHER OUTCOMES:
Exploratory outcome-Proportion and location of different immune cell subsets at baseline and during treatment associated with cCR or near cCR | From baseline to withdrawal of consent or death (whichever occurs first), up to 8 years
  Proportion and location of different immune cell subsets will be assessed by single-cell sequencing, immunohistochemistry, and multiplex fluorescence immunohistochemistry.
Exploratory outcome-Tumor gene alterations associated with cCR or near cCR | From baseline to withdrawal of consent or death (whichever occurs first), up to 8 years
  Tumor gene alterations will be assessed by whole exome sequencing using tissue or blood samples.
Exploratory outcome-Baseline clinical and pathological characteristics associated with cCR or near cCR | From baseline to withdrawal of consent or death (whichever occurs first), up to 8 years
  Baseline clinical characteristics include age of onset, gender, family history, pathological type of tumor, primary tumor site, tumor size, and previous treatment.
Exploratory outcome-Baseline and longitudinal on-treatment MR image characteristics associated with cCR or near cCR | From baseline to withdrawal of consent or death (whichever occurs first), up to 8 years
  MR image characteristics at baseline and their changes when tumor responded or progressed

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No